CLINICAL TRIAL: NCT01361477
Title: Data Registry of ICU Siamitra and ICU Salad-Samung
Brief Title: Data Registry of Intensive Care Unit (ICU) Siamitra and Intensive Care Unit (ICU) Salad-Samung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suneerat Kongsayreepong, MD, Professor, Mahidol University
Other Study IDs: Si227/2011
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Complication
Keywords: General surgical ICU; ICU Siamitra; ICU Salad-Samung; Data registry; ICU refusal; ICU complications; ICU resource utilization; Adverse events; ICU readmission; intraoperative hypotension; intraoperative cardiac arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient: 1. Prolonged ICU stay
  2. Unplanned ICU admission
  3. Complication/adversel during ICU admission
  4. Result of intraoperative complications and admission to ICU 5 Result of early postoperative (within 7 days) and ICU admission

SUMMARY:
As a general surgical intensive care units of the biggest tertiary referral university of Thailand with more than 1,000 admissions/year, recently, more complicated perioperative care surgical patients were accepted with high complications, morbidities, mortality and resource utilization. Good data registration was needed to provide information for quality improvement and resource allocation. This prospective observational (crosssectional) study was designed to register patient > 18 years who will be admitted to these ICUs to explore the adequacy of these ICUs services, resource utilization (ICU length of stay and ventilator day), ICU complications, adverse outcome /ICU readmission within 72 hours after discharging from ICU. In addition, severe hemodynamic, respiratory, or neurological disturbance or complication intra and early postoperative (within 7 days after operation) that lead to ICU admission eg, intraoperative hypotension, intraoperative cardiac arrest, perioperative pulmonary aspirtaion will also be studied.

DETAILED DESCRIPTION:
This prospective obseverational study wae ans will be done in all surgical patient (age . 18 yeras) admitted to the general surgical ICU (ICU Siammitra and ICU Salad-sumang) of the Department of Anesthesiology, Siriraj Hospital, Faculty of Medicine, Mahidol UNiversity, Bangkok, Thailand. After approval by the IRB of Siriaj Hospital, all information of the patients admiited to the ICUs were carefully recorded included patient demographic data, comorbidities, type of anesthesia, type of surgery, complication associated with anesthesia and surgery, type of ICU admission and course in ICU including outcome as Iresouce utilization (cost in ICU, ventilator day, ICU and hosital length of stay. Morbidity occcuring in ICU, 28 and 90 days mortality also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Surgical patients

Exclusion Criteria:

* Patient undergoing cardiothoracic surgery, traumatic surgery, neurosurgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (> 18 years), admitting to ICU Siamitra and ICU Salad-Samung
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-05 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Prolonged ICU stay | 9 years
  Incidence and factors associated with prolonged ICU stay

SECONDARY OUTCOMES:
ICU complication, resource utilization and adverse events/ICU readmission within 72 hours after discharging from ICU | 9 years
  ICU complication, resource utilization and adverse events/ICU admission within 72 hours after discharging from ICU
Unplanned ICU admission | 9 years
  All unplanned ICU Admission (from OR and from floor)
outcome of complications occurring intraoperative and admitting to ICU | 9 years
  all complication including: intraoperative cardiac arrest, hypotension
sepsis and septic shock on ICU admission | 9 years
  incidence, clinical course and outcome of surgical septic shock admitting to ICU

CONTACTS AND LOCATIONS:
Overall Officials: Suneerat Kongsereepong, MD, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - ICU Siamitra and ICU Salad-Samung, Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok
  - ICU Siamitra and ICU Salad-Samung, Siriraj Hospital, Bangkoknoi, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Capuzzo M, Moreno RP, Alvisi R. Admission and discharge of critically ill patients. Curr Opin Crit Care. 2010 Oct;16(5):499-504. doi: 10.1097/MCC.0b013e32833cb874. PMID 20644469